CLINICAL TRIAL: NCT03544697
Title: Easy Way of Choosing Rectangular Expander and Getting Maximum Benefit From Expanded Tissue
Status: Completed | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ersin Aksam, Assistant Professor, Izmir Katip Celebi University
Other Study IDs: IzmirKCU-Plastik1
Record Dates: First submitted 2018-05-21; First posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Burn Scar; Scalp Wound
MeSH Terms: interventions — Wound Healing; Surgical Flaps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Skin expansion and repair with flaps: The tissue expander was inserted into the scalp in 17 patients and supraclavicular area in two patients.
  Interventions: Procedure: Skin expansion and repair with flaps

INTERVENTIONS:
Procedure: Skin expansion and repair with flaps

SUMMARY:
Background: Tissue expanders are widely used for reconstruction of tissue defects. The choice of expander and planning the flap is complicated for the inexperienced surgeon.

Objective: To demonstrate the choice of expander sizes proper for the tissue defect and maximum advancement technique during the defect coverage.

Methods: The present study included 19 patients who were operated between January 2013 and January 2017. The expander projection was chosen in the manner that it would be more than the half length of the defect to be occurred and the expander width was chosen as wide as possible based on the area of its placement. After the expansion was completed, advancement method was used to cover the defect.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with rectangular tissue expanders.
* Patients who attended to at least postoperative six months control.

Exclusion Criteria:

* Patients treated with tissue expanders other than rectangular expanders.
* Patients who did not attend to postoperative controls.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The present study included 19 patients who were operated using one rectangular expander between January 2013 and January 2017.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Scar revision | 6 months
  Closure of defect

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] NEUMANN CG. The expansion of an area of skin by progressive distention of a subcutaneous balloon; use of the method for securing skin for subtotal reconstruction of the ear. Plast Reconstr Surg (1946). 1957 Feb;19(2):124-30. doi: 10.1097/00006534-195702000-00004. No abstract available. PMID 13419574
- [Background] Radovan C. Breast reconstruction after mastectomy using the temporary expander. Plast Reconstr Surg. 1982 Feb;69(2):195-208. doi: 10.1097/00006534-198202000-00001. PMID 7054790
- [Background] Pamplona DC, Velloso RQ, Radwanski HN. On skin expansion. J Mech Behav Biomed Mater. 2014 Jan;29:655-62. doi: 10.1016/j.jmbbm.2013.03.023. Epub 2013 Apr 19. PMID 23651568
- [Background] Radovan C. Tissue expansion in soft-tissue reconstruction. Plast Reconstr Surg. 1984 Oct;74(4):482-92. doi: 10.1097/00006534-198410000-00005. PMID 6484035
- [Background] Manders EK, Schenden MJ, Furrey JA, Hetzler PT, Davis TS, Graham WP 3rd. Soft-tissue expansion: concepts and complications. Plast Reconstr Surg. 1984 Oct;74(4):493-507. doi: 10.1097/00006534-198410000-00007. PMID 6484036
- [Background] Hudson DA. Maximising the use of tissue expanded flaps. Br J Plast Surg. 2003 Dec;56(8):784-90. doi: 10.1016/s0007-1226(03)00379-5. PMID 14615253
- [Background] Pamplona DC, Weber HI, Leta FR. Optimization of the use of skin expanders. Skin Res Technol. 2014 Nov;20(4):463-72. doi: 10.1111/srt.12141. Epub 2014 Feb 17. PMID 24527999
- [Background] Kiyokawa K, Rikimaru H, Inoue Y, Tai Y. A new concept and technique for reconstructing skin defects in the cheek region: an unfolded cube advancement flap. Plast Reconstr Surg. 2004 Mar;113(3):985-91. doi: 10.1097/01.prs.0000105045.57704.44. No abstract available. PMID 15108895
- [Background] Ueda K, Hara M, Okada M, Kurokawa N, Otani K, Nuri T. Lambda incision for effective tissue expansion. J Plast Reconstr Aesthet Surg. 2010 Oct;63(10):1682-7. doi: 10.1016/j.bjps.2009.09.015. Epub 2009 Nov 11. PMID 19906567
- [Background] Yenidunya MO. The bi-lobed flap design on expanded skin of the face and neck region. Plast Reconstr Surg. 1998 May;101(6):1741-2. doi: 10.1097/00006534-199805000-00066. No abstract available. PMID 9583521